CLINICAL TRIAL: NCT06737016
Title: Efficacy and Safety of Tamsulosin, a Selective Alpha-1 Adrenergic Blocker, for Children with Posterior Urethral Valve: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Tamsulosin for Children with Posterior Urethral Valve.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tamsulosin & PUV
Record Dates: First submitted 2024-11-29; First posted 2024-12-17 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Posterior Urethral Valve
Keywords: Posterior Urethral Valve
MeSH Terms: interventions — Tamsulosin; oxybutynin; Trimethoprim; Sulfamethoxazole

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxybutynin and Trimethoprim/sulphamethoxazole (Active Comparator): Patients will undergo maintenance therapy Anticholinergic, oxybutynin and Continous Antibiotic Prophylaxis,Trimethoprim/sulphamethoxazole daily
  Interventions: Drug: Oxybutynin; Drug: Trimethoprim/sulfamethoxazole (TMP/SMZ)
- Tamsulosin, Oxybutynin and Trimethoprim/sulfamethoxazole (Experimental): Patients will undergo maintenance therapy Tamsulosin in addition to Anticholinergic, Oxybutynin and Continous Antibiotic Prophylaxis, Trimethoprim/sulfamethoxazole daily
  Interventions: Drug: Tamsulosin; Drug: Oxybutynin; Drug: Trimethoprim/sulfamethoxazole (TMP/SMZ)

INTERVENTIONS:
Drug: Tamsulosin — Children will be maintained on an oral dose of Tamsulosin 0.1 mg once daily (in children aged less than 2 years old) and 0.2 mg once daily (≥2 years old).
  Arms: Tamsulosin, Oxybutynin and Trimethoprim/sulfamethoxazole
Drug: Oxybutynin — Children will be maintained on an oral dose of Oxybutynin 0.2 mg/kg 2 times daily.
Drug: Trimethoprim/sulfamethoxazole (TMP/SMZ) — Children will be maintained on an oral prophylactic dose of Trimethoprim/sulfamethoxazole 2 mg/kg single dose at night.

SUMMARY:
To determine whether there is a role for Tamsulosin, A Selective Alpha-1 Adrenergic Blocker, as therapy in children with Posterior Urethral Valve post valve ablation , and whether there are side effects involved.

DETAILED DESCRIPTION:
We aim to evaluate the safety and efficacy of alpha adrenergic blocker, tamsulosin, in children with posterior urethral valves regarding:

* Effect on upper urinary tract (Hydronephrosis improvement, Vesicoureteric Reflux resolution and renal function)
* Effect on bladder outlet resistance
* Effect on intravesical detrusor pressure
* Febrile Urinary Tract Infection recurrence

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of PUV.

Exclusion Criteria:

1. Patients with other conditions that can potentially affect lower or upper urinary tract functions (e.g. spinal dysraphism, anorectal malformation and prune belly syndrome)
2. Patients who were treated with urinary diversion as vesicostomy or cutaneous ureterostomy.
3. Patients who had primary treatment of PUV ablation at other hospitals.
4. Contraindications to α blocker treatment.
5. Patients who refuse to participate in the study

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The effect of alpha adrenergic blocker, tamsulosin, on upper urinary tract in children with posterior urethral valves. | 1 year
  The effect of alpha adrenergic blocker, tamsulosin, on upper urinary tract in children with posterior urethral valves. This will be assessed by:
  - Change in Hydronephrosis grading (resolution of low grade (I or II) Hydronephrosis or downgrading of high grade (III or IV) Hydronephrosis to grade II or less)
The safety of alpha adrenergic blocker, tamsulosin, in children with posterior urethral valves. | 1 year
  Number of children with treatment related adverse effects. Potential side effects will be discussed after initiating therapy, including postural hypotension, dizziness, headache and rhinitis.

SECONDARY OUTCOMES:
The effect of alpha adrenergic blocker, tamsulosin, on lower urinary tract in children with posterior urethral valves. | 1 year
  The effect of alpha adrenergic blocker, tamsulosin, on lower urinary tract in children with posterior urethral valves.
  This will be assessed by:
  • Change in Bladder neck Hypertrophy ( as determined by Voiding Cysto-Urethrogram imaging)
Febrile Urinary Tract Infections recurrence | 1 year
  fever 38.5C or higher with a positive urinalysis and bacterial growth

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Tarek Hafez, Study Chair — Urology and Nephrology center,Mansoura university; Tamer Helmy, Study Director — Urology and Nephrology center,Mansoura university; Ahmed Elkashef, Study Director — Urology and Nephrology center,Mansoura university; Mohamed Hussiny, Principal Investigator — Urology and Nephrology center,Mansoura university
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin PF, Homsy YL, Masel JL, Cain MP, Casale AJ, Rink RC. alpha-Adrenergic blockade in children with neuropathic and nonneuropathic voiding dysfunction. J Urol. 1999 Sep;162(3 Pt 2):1064-7. doi: 10.1016/S0022-5347(01)68067-4. PMID 10458432
- [Background] Abraham MK, Nasir AR, Sudarsanan B, Puzhankara R, Kedari PM, Unnithan GR, Damisetti KR, Narayanan T. Role of alpha adrenergic blocker in the management of posterior urethral valves. Pediatr Surg Int. 2009 Dec;25(12):1113-5. doi: 10.1007/s00383-009-2469-9. Epub 2009 Sep 1. PMID 19727771